CLINICAL TRIAL: NCT07252856
Title: CrOss-cultural Model for Postdischarge Assistance and Sustainable Digital Solutions in Phase III Cardiac Rehabilitation: a Randomized Controlled Trial
Brief Title: Transcultural Digital Solutions in Phase III Cardiac Rehabilitation
Acronym: COMPASS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COMPASS
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Myocardial Infarction
MeSH Terms: conditions — Heart Failure; Myocardial Infarction | interventions — AT1G72490 protein, Arabidopsis

STUDY DESIGN:
Intervention Model Description: Randomized Type I hybrid study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEEPER (Experimental): As "Standard Care" plus every 15 days in the first month and at least once a month chat with healthcare professional that will keep posted with the patient and the staff (nurse, physiotherapist, cardiologist) for all the issues raised by the patients. chat with answer within 72 hours. Graphical medicine to increase patients' awareness.
  Interventions: Behavioral: DEEPER
- Standard of care (No Intervention): Discharge after phase II, LC9 evaluation, discharge indications, website indication for every country language support (from the European Society of Preventive Cardiology). FU contact by phone at 3 months, clinical visit at 6 months [6 month LE9 assessment (primary endpoint)] and contact by phone at 1 year for MACE evaluation.

INTERVENTIONS:
Behavioral: DEEPER — A transcultural scientific digital platform (Rehab companion, Inselspital, University Hospital of Bern) for content delivery, feedback and digital biomarker monitoring will be made available.
  Arms: DEEPER

SUMMARY:
Multicenter Prospective Controlled Randomized Trial, open-label, in patients with atherosclerotic cardiovascular disease (ASCVD) (acute coronary syndrome or chronic coronary syndrome and ischemic heart failure) and an approved indication for cardiac rehabilitation (CR). Patients completing phase II CR will be randomized 1:1 to usual Phase-III care (standard care) versus standard care plus the Digitally-Enhanced Extended PrEvention & Rehabilitation (DEEPER) package (intervention). Primary outcome is 6-month change in composite Life's Crucial 9 (LC9) (LE8 + PHQ-9).

DETAILED DESCRIPTION:
Multicenter Prospective Controlled Randomized Trial, open-label, in patients with atherosclerotic cardiovascular disease (ASCVD) (acute coronary syndrome or chronic coronary syndrome and ischemic heart failure) and an approved indication for cardiac rehabilitation (CR). Patients completing phase II CR will be randomized 1:1 to usual Phase-III care (standard care) versus standard care plus the Digitally-Enhanced Extended PrEvention & Rehabilitation (DEEPER) package (intervention). Primary outcome is 6-month change in composite Life's Crucial 9 (LE9) (LE8 + PHQ-9). Intervention (DEEPER) will include informative modules (patient will choose among graphic medicine, video or interactive messaging) that will be delivered every two weeks via secure digital platform (or booklet if offline); monthly motivational messages; moderated peer-support forum with leaderboard; remote wearable step/sleep upload with personalized content assignment and feedback, linked to the hospital interactive digital platform (Rehab companion).

Patients will be encouraged to have their own device to be adopted as lifelong maintenance. Nevertheless, centres will provide a smartwatch (fitbit) to all the patients enrolled in the trial as incentive for study participation and to uniformly collect study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, men and women;
* patients with atherosclerotic cardiovascular disease (ASCVD) (acute coronary syndrome or chronic coronary syndrome and ischemic heart failure);
* patients who completed phase II CR and are therefore eligible for CR phase III (maintenance).

Exclusion Criteria:

* Unable to sign the informed consent;
* unable or unwilling to use digital devices due to mental/cognitive issues or without a support person helping them to access the respective technical devices;
* pregnant, lactating or women planning pregnancy during the course of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2026-04-05 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
6-month change in composite Life's Essential 9 (LE9) | 6-month change
  LC9 is defined by the American Heart Association's Life's Essential 8 (LE8), complemented by the Patient Health Questionnaire (PHQ-9), collectively referred to as "LC9 [blood pressure, non-high-density lipoprotein cholesterol (HDL), diet questionnaire, physical activity, smoking habits, sleep health, body mass index (BMI), hemoglobin A1c (HbA1c, %), PHQ9 from questionnaire).

SECONDARY OUTCOMES:
Individual LE8 sub-scores | 6-month change
  Reported as differences in the absolute value among the two groups (median and (IQR)
Major adverse cardiovascular event (MACE) | 6 months
  defined as a composite of death of any cause, myocardial infarction, unplanned revascularization, rehospitalization for any cause, stroke, considered in a hierarchical way and as single endpoint
Major adverse cardiovascular event (MACE) | 1 year
  defined as a composite of death of any cause, myocardial infarction, unplanned revascularization, rehospitalization for any cause, stroke, considered in a hierarchical way and as single endpoint
GAD 7 | Changes between baseline and 6-month follow-up
  anxiety score; Seven-item questionnaire that assesses the severity of anxiety symptoms over the past two weeks, with a total score ranging from 0 to 21
PHQ 9 | Changes between baseline and 6-month follow-up
  depression score; The PHQ-9 score ranges from 0 to 27. Scores between 5 and 9 indicate the presence of subthreshold depression.
Physical fitness | Changes between baseline and 6-month follow-up
  distance achieved in 6-minute walking test
VO2 peak | Changes between baseline and 6-month follow-up
  cardiopulmonary test (CPET)
30 second sit-to -stand test | Changes between baseline and 6-month follow-up
  number of times the patient stands in 30 seconds
Hand-grip strength | Changes between baseline and 6-month follow-up
  maximum voluntary muscle strength measured by dynamometer
Steps per day | Changes between baseline and 6-month follow-up
  amount of steps during the day
Waist circumference | Changes between baseline and 6-month follow-up
  Waist circumference in cm
counter movement jump test. | Changes between baseline and 6-month follow-up
  Maximum power measured by dynamometer; difference in the absolute value among the two groups
Compliance with study treatment | 6 months
  Compliance with study treatment defined as number (percentage) of patients who will attend the sessions provided and will complete the study.
Economic impact of the CR pathways and financial sustainability: standard care versus stardard care plus the DEEPER package | 6 months
  Direct costs of the two pathways, estimated using Activity Based Costing and financial sustainability measured with a budget impact analysis (BIA). Results reported as mean difference and standard deviation (SD) between groups.
  Cost per patient and cost-effectiveness ratio will be calculated per group of treatment.
Acceptance of the usual care and the DEEPER package pathway using the Service User Technology Acceptance Questionnaire (SUTAQ) average values | 6 months
  Responses to SUTAQ-based questionnaire administered to patients involved in the study, analyzed through a seven items scale scoring. Results reported as mean, p-value and linear regression models for enhanced care, increased accessibility, privacy and discomfort, care personnel concerns, telerehabilitation as substitution and satisfaction.
Assessment of social, ethical and equity dimensions. | 6 months
  Perceptions reported by the patients, measured with a seven item Likert scale structured questionnaire based on the EUnetHTA Core Model dimensions, comparing standard care versus DEEPER package (mean and p-value)
Social costs | 6 months
  Analysis of the indirect and out of pocket costs as average value in case of standard care and DEEPER package, to define the social costs related to the interventions.
Safety endpoint | 6 months
  Musculo-skeletal injuries (requiring medical attention) and Arrhythmias (atrial fibrillation, supraventricular tachycardia, ventricular tachycardia) requiring medical attention and an emergency room or ambulatory visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nuccia Morici, MD, Principal Investigator — IRCCS Fondazione Don Gnocchi
Locations (5):
- KU Leuven, Kaatje Goetschalckx, KU Leuven, Leuven, Belgium
- Italy (2):
  - Carlo Cattaneo - LIUC University, Castellanza
  - Istituti Clinici Scientifici Maugeri SpA - Società Benefit, IRCCS, Lumezzane, Lumezzane
- Associação para Investigação e Desenvolvimento da Faculdade de Medicina - AIDFM, representing Instituto Medicina Preventiva e Saúde Public (IMPSP) & Instituto de Saúde Ambiental (ISAMB), Lisbon, Portugal
- Centre for Rehabilitation & Sports Medicine, Inselspital, University Hospital of Bern, Bern Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
COMPASS research outputs will be primarily disseminated through the Zenodo repository to guarantee persistent access. To enhance discoverability, we will implement a FAIR Data Point following the official FDP specification, initially through a self-hosted solution during the active project phase. As the ecosystem evolves, we plan to migrate this functionality to established platforms like FAIR sharing, contingent on their ability to fully support our metadata requirements for cardiac rehabilitation data.
Supporting Information: Study Protocol, SAP
Time Frame: After the study completion
Access Criteria: Data anonymization process